CLINICAL TRIAL: NCT00358072
Title: Treatment of Adult Acute Lymphoblastic Leukemia Using a Post-remission Programme Whose Intensity Varies Depending on the Risk Class Defined on the Basis of Minimal Residual Disease.
Brief Title: Treatment of Adult ALL With an MRD-directed Programme.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northern Italy Leukemia Group (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Renato Bassan, MD, Ospedali Riuniti, Div. Ematologia, Bergamo, Italy
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NILG-ALL 09/00
Record Dates: First submitted 2006-07-26; First posted 2006-07-28 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute lymphoblastic leukemia; Adult patients; Minimal residual disease; Risk-oriented therapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Application of combination chemotherapy aimed to reduce MRD burden in unselected patients, followed by MRD-adjusted therapy that range from maintenance chemotherapy (MRD-negative patients) to allogeneic SCT (MRD-positive patients) or high-dose therapy with autologous blood stem cell support (MRD-positive patients without compatible donor for allogeneic SCT)
  Interventions: Behavioral: Postremission consolidation based on MRD status

INTERVENTIONS:
Behavioral: Postremission consolidation based on MRD status — Application of combination chemotherapy aimed to reduce MRD burden in unselected patients, followed by MRD-adjusted therapy that range from maintenance chemotherapy (MRD-negative patients) to allogeneic SCT (MRD-positive patients) or high-dose therapy with autologous blood stem cell support (MRD-positive patients without compatible donor for allogeneic SCT)
  Other Names: MRD-guided therapy

SUMMARY:
The study aims to optimize the concept of risk-oriented postremission consolidation therapy, by offering (i) standard consolidation-maintenance to patients at lowest risk of relapse as defined by MRD(Minimal Residual Disease) negative status, and (ii) allogeneic stem cell transplantation (related/unrelated donor available) or multicycle high-dose therapy with autologous blood stem cell transplant (no donor) to patients at highest risk of relapse as defined by MRD+ status.

The prognostic role of MRD evaluation in unselected patients will be evaluated.

DETAILED DESCRIPTION:
Improved outcome of adult ALL through the application of:

* Risk-adapted induction (cycle no. 1: IVAP i.e idarubicin-vincristine-asparaginase-prednisone, plus fractionated cyclophosphamide in T-ALL,and imatinib in Ph/BCR-ABL+ ALL)
* Risk stratification (clinical) according to morphology, immunophenotype, cytogentics and molecular biology results. Standard risk (SR) is defined by pre-B CD10+ phenotype, Ph/BCR-ABL- status, and a blast count <10x10e9/L. All other subgroups are HR (high-risk) except for Ph/BCR-ABL+ and t(4;11)+ ALL (VHR, very high-risk)
* Homogeneous early consolidation programme including both conventional therapy with idarubicin-vincristine-cyclophosphamide-dexamethasone/prednisone(cycles no. 2,3,5,6,8) and high-dose treatemt with MTX/Ara-C (cycles no. 4,7) and meningeal prophylaxis (triple intrathecal therapy x8-12, skull irradiation), plus imatinib in Ph+ ALL (Phase A). Autologous bllo stem cells are mobilized and cryopreserved after cycle no. 4.
* Serial evaluation of minimal residual disease (MRD) with RQ-PCT technology, aiming to define in individual patients the rate of reduction during early consolidation. The molecular study was centralized and aimed at obtaining one or more patient-specific probe(s)with a sensitivity of at least 10e-3. Patient bone marrow was sampled for MRD analysis at timepoints 13 i.e. after cycles no.3,5, and 7. Only patients with a negative result at timepoint 3 and a negative/low positive (<10e-4) result at timepoint 3 are considered MRD-, all other combinations being regarded MRD+.
* Phase B therapy according to MRD results and ALL subset:

  * MRD- nonPh/t(4;11): standard maintenance
  * MRD+ nonPh/t(4;11): allogeneic stem cell transplantation (from sibling/MUD) or, alternatively, intensified high-dose therapy (2-4 "hypercycles")with autologous stem cell support and anti CD20 MoAb (if CD20+), followed by maintenance. Each "hypercycle" consists of high-dose mercaptopurine-etoposide-melphalan (cycles no. 1,3) or methotrexate-cytarabine (cycles no. 2,4)
  * MRD unknown nonPh/t(4;11): treatment by clinical risk (SR: maintenance; HR, as per MRD+)
  * Ph/t(4;11)+: allogeneic stem cell transplantation as soon as possible into complete remission; if a transplant is not possible, consolidation is as for HR patients. each cycle is supplemented by imatinib in Ph+ ALL

The illustrated strategy aims to optimize postremission consolidation therapy by offering standard treatment "only" to patients at lowest risk of relapse (MRD-), thereby reducing the risks of high dose treatments (expected TRM from allogeneic SCT 20-30%), while maintaining the latter approach in MRD+ cases and very HR subsets.

The prognostic role of MRD evaluation in unselected patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Untreated Acute lymphoblastic leukemia or lymphoblastic lymphoma (T-cell, precursor B-cell)
* Age 15-65 years (older patients if biologically fit according to responsible physician)
* Written informed consent

Exclusion Criteria:

* Any co-morbidity precluding the administration of intensive chemotherapy for adult ALL

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2000-05; Primary Completion 2006-12 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Disease-free survival at 5 years | 5 year from date of complete remission

SECONDARY OUTCOMES:
Complete remission | 4 or 8 weeks from date of therapy start
Overall survival | 5 years from date of diagnosis
Cumulative incidence of relpase | 5 years from date of complete remission
Remissional deaths | 4 weeks from date of therapy start
Nonlethal toxicity | 5 years from date of therapy start

CONTACTS AND LOCATIONS:
Overall Officials: Bassan Renato, MD, Principal Investigator — Azienda Ospedaliera Ospedali Riuniti di Bergamo
Locations (15):
- Italy (15):
  - Ospedali Riuniti di Bergamo, Bergamo, BG
  - Divisione Ematologia Spedali Civili, Brescia, BS
  - Divisione di Ematologia e TMO Ospedale San Maurizio, Bolzano, BZ
  - U.O. Ematologia e Centro TMO Ospedale Armando Businco, Cagliari, CA
  - Ematologia Azienda Ospedaliera S.Croce e Carle, Cuneo, CN
  - U.S. Ematologia - Centro TMO Istituti Ospedalieri, Cremona, CR
  - Ematologia AOU Careggi, Florence, FI
  - Ematologia Centro TMO Fondazione IRCSS Ospedale Maggiore, Milan, MI
  - Ematologia e TMO Ospedale San Raffaele, Milan, MI
  - Ematologia - TMO Ospedale San Gerardo, Monza, MI
  - Oncoematologia e TMO Dipartimento Oncologico, Palermo, PA
  - Ematologia 2 Ospedale San Giovanni Battista, Torino, TO
  - Divisione Ematologia Ospedale Umberto I, Mestre, VE
  - Oncologia ed Ematologia Oncologica Institution Regione Veneto, ULSS n.13 - Presidi Ospedalieri di Noale, Mirano, Dolo, Noale, VE
  - Ematologia Ospedale San Bortolo, Vicenza, VI

REFERENCES:
- [Result] Bassan R, Spinelli O, Oldani e et al. Minimal residual disease (MRD) and risk-oriented therapy in adult acute lymhoblastic leukemia (ALL). Blood (ASH Annual Meeting Abstract) 106: abstract 1836, 2005.
- [Result] Bassan R, Spinelli O, Oldani E, Intermesoli T, Tosi M, Peruta B, Rossi G, Borlenghi E, Pogliani EM, Terruzzi E, Fabris P, Cassibba V, Lambertenghi-Deliliers G, Cortelezzi A, Bosi A, Gianfaldoni G, Ciceri F, Bernardi M, Gallamini A, Mattei D, Di Bona E, Romani C, Scattolin AM, Barbui T, Rambaldi A. Improved risk classification for risk-specific therapy based on the molecular study of minimal residual disease (MRD) in adult acute lymphoblastic leukemia (ALL). Blood. 2009 Apr 30;113(18):4153-62. doi: 10.1182/blood-2008-11-185132. Epub 2009 Jan 13. PMID 19141862
- [Result] Bassan R, Rossi G, Pogliani EM, Di Bona E, Angelucci E, Cavattoni I, Lambertenghi-Deliliers G, Mannelli F, Levis A, Ciceri F, Mattei D, Borlenghi E, Terruzzi E, Borghero C, Romani C, Spinelli O, Tosi M, Oldani E, Intermesoli T, Rambaldi A. Chemotherapy-phased imatinib pulses improve long-term outcome of adult patients with Philadelphia chromosome-positive acute lymphoblastic leukemia: Northern Italy Leukemia Group protocol 09/00. J Clin Oncol. 2010 Aug 1;28(22):3644-52. doi: 10.1200/JCO.2010.28.1287. Epub 2010 Jul 6. PMID 20606084
- [Derived] Mannelli F, Gianfaldoni G, Intermesoli T, Cattaneo C, Borlenghi E, Cortelazzo S, Cavattoni I, Pogliani EM, Fumagalli M, Angelucci E, Romani C, Ciceri F, Corti C, Scattolin A, Cortelezzi A, Mattei D, Audisio E, Spinelli O, Oldani E, Bosi A, Rambaldi A, Bassan R. CD20 expression has no prognostic role in Philadelphia-negative B-precursor acute lymphoblastic leukemia: new insights from the molecular study of minimal residual disease. Haematologica. 2012 Apr;97(4):568-71. doi: 10.3324/haematol.2011.054064. Epub 2011 Nov 4. PMID 22058217